CLINICAL TRIAL: NCT02917824
Title: Intensity, Specificity and Reversibility of Inspiratory Muscle Training in Asthmatics: a Randomized Clinical Trial
Brief Title: Intensity, Specificity and Reversibility of Inspiratory Muscle Training in Asthmatics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal do Rio Grande do Norte (Other)
Responsible Party: Principal Investigator, Gardenia Maria Holanda Ferreira, Principal Investigator, Universidade Federal do Rio Grande do Norte
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1.533.228
Record Dates: First submitted 2016-09-25; First posted 2016-09-28 (Estimated); Last update posted 2019-09-10 (Actual); Status verified 2019-09

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-intensity IMT (Experimental): Participants enrolled in this arm received high-intensity IMT
  Interventions: Device: High-intensity IMT
- Low-intensity IMT (Active Comparator): Participants enrolled in this arm received low-intensity IMT
  Interventions: Device: Low-intensity IMT

INTERVENTIONS:
Device: High-intensity IMT — 30 breaths at 50% of the maximal inspiratory pressure, twice daily for 6 weeks
  Arms: High-intensity IMT
Device: Low-intensity IMT — 30 breaths at 15% of the maximal inspiratory pressure, twice daily for 6 weeks
  Arms: Low-intensity IMT

SUMMARY:
Inspiratory muscle training (IMT) can reverse or delay the complications from the deterioration of inspiratory muscle function in asthma. Thus, the IMT has been considered a treatment option for people with asthma. The aim of this study is to investigate the training principles of intensity, specificity and reversibility of IMT in asthmatics.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of asthma
* Adults (18 - 60 years)

Exclusion Criteria:

* Inability to perform the protocol established by the study
* Others respiratory diseases
* Request for study withdrawal

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Change in inspiratory muscle strength | Baseline, 6 weeks later and 6 weeks after training
  Maximal inspiratory pressure
Change in expiratory muscle strength | Baseline, 6 weeks later and 6 weeks after training
  Maximal expiratory pressure

SECONDARY OUTCOMES:
Change in asthma control | Baseline, 6 weeks later and 6 weeks after training
  Asthma Control Questionnaire measures the adequacy of asthma control and change in asthma control which occurs either spontaneously or as a result of treatment. Scores range between 0 (totally controlled) and 6 (severely uncontrolled)
Change in quality of life | Baseline, 6 weeks later and 6 weeks after training
  Asthma Quality of Life Questionnaire is a disease-specific health-related quality of life instrument that taps both physical and emotional impact of disease. Scores range 1-7, with higher scores indicating better quality of life.
Change in six minute walk test distance | Baseline, 6 weeks later and 6 weeks after training
  Six-minute walk test (6MWT)
Change in forced vital capacity | Baseline, 6 weeks later and 6 weeks after training
  Forced vital capacity in litres and % of predicted
Change in forced expiratory volume | Baseline, 6 weeks later and 6 weeks after training
  Forced expiratory volume in litres and % of predicted
Change in forced expiratory volume/forced vital capacity | Baseline, 6 weeks later and 6 weeks after training
  Forced expiratory volume/forced vital capacity
Change in inspiratory muscle activity | Baseline, 6 weeks later and 6 weeks after training
  Surface electromyography of inspiratory muscles

CONTACTS AND LOCATIONS:
Locations (1):
- Gardenia Maria Holanda Ferreira, Natal, Rio Grande do Norte, Brazil